CLINICAL TRIAL: NCT03177330
Title: Safety and Efficacy of Heparin Dosing Score Protocol for Anticoagulation During Polymyxin-B Hemoperfusion: a Retrospective Study
Brief Title: Safety and Efficacy of Heparin Dosing Score Protocol for Polymyxin-B Hemoperfusion
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201704033RIND
Record Dates: First submitted 2017-06-04; First posted 2017-06-06 (Actual); Last update posted 2017-06-06 (Actual); Status verified 2017-06

CONDITIONS: Septic Shock; Polymyxin B Hemoperfusion
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Polymyxin B hemoperfusion (PMX-HP) is mainly used to remove endotoxins in septic shock patients with intra-abdominal infections. Because of the concerns of postoperative bleeding, physicians may hesitate to use anticoagulation in patients with septic shock within a few hours after an abdominal operation. We developed a heparin dosing score protocol for heparin dosage adjustment. The purpose of the study is to examine the safety and efficacy of the heparin dosing score protocol.

ELIGIBILITY:
Inclusion Criteria:

* intra-abdominal septic shock patients or documented Gram-negative bacterial septic shock patients who received polymyxin-B hemoperfusion in National Taiwan University Hospital during October 2013-December 2016

Exclusion Criteria:

* pregnant woman
* patients with do-not-resuscitate declaration
* uncontrolled bleeding within 24hr

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: intra-abdominal septic shock patients or documented Gram-negative bacterial septic shock patients who received polymyxin-B hemoperfusion
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2017-05-15 (Actual); Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
premature cartridge clotting rate | 2 hours
  the incidence of premature cartridge clotting within 2hr

SECONDARY OUTCOMES:
bleeding event rate | 24 hours
  the incidence of substantial bleeding event within 24hr

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology, NTUH, Taipei, Taiwan, Taipei, Taiwan